CLINICAL TRIAL: NCT04238013
Title: Influence of Whole Body Vibration on Neuromodulation of Ankle Muscles in Persons With SCI
Brief Title: Neuromodulation of Ankle Muscles in Persons With SCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the ongoing COVID-19 pandemic, my recruitment progress was delayed to the point that I had to reevaluate the feasibility of continuing data collection.
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Edelle Field-Fote, PT, PhD, Director, Spinal Injury Research & The Hulse Spinal Injury Laboratory, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 777; F31HD101151 (NIH)
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Spinal Cord Injuries; Spastic Gait; Foot Drop
MeSH Terms: conditions — Spinal Cord Injuries; Gait Disorders, Neurologic; Peroneal Neuropathies | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticospinal Tract Excitability (Active Comparator): During the Corticospinal Tract Excitability arm, corticospinal excitability will be assessed by measuring motor evoked potentials after transcranial magnetic stimulation pre-post each intervention in conjunction with other outcome measures.
  Interventions: Other: Whole Body Vibration (WBV); Other: Electrical Stimulation
- Spinal Reflex Circuit Excitability (Active Comparator): During the Spinal Reflex Circuit Excitability arm, spinal reflex circuit excitability will be assessed by measuring low frequency depression after Hoffmann-Reflex testing pre-post each intervention in conjunction with other outcome measures.
  Interventions: Other: Whole Body Vibration (WBV); Other: Electrical Stimulation

INTERVENTIONS:
Other: Whole Body Vibration (WBV) — The WBV session will consist of 8 bouts of 45s vibration (50Hz) with a minute of rest in between each bout.
Other: Electrical Stimulation — The electrical stimulation intervention serves to account for any effects of standing and/or of repeated performance of the sit-to-stand behavior on neurophysiological outcomes. In the electrical stimulation intervention, participants will receive electrical stimulation while standing on the vibration platform for 8 bouts for 45s with a minute of rest in between without vibration.

SUMMARY:
The ability to voluntarily move the ankles is important for walking. After spinal cord injury (SCI), this ability is impaired because of changes in the communication between the brain, spinal cord, and body. Whole body vibration (WBV) is a treatment that increases voluntary muscle control and decreases uncontrollable muscle movement in people with SCI. The purpose of this study is to understand how WBV can impact ankle control and uncontrollable muscle movement.

DETAILED DESCRIPTION:
Spinal cord injury can result in impaired walking ability and decreased independence in daily activities such as standing and transfers. The ability to voluntarily control the ankle muscles is an important component of walking that is impacted by changes in the corticospinal tract and the spinal reflex circuits. These changes have been associated with the inability to dorsiflex the ankle during swing phase (foot drop) and uncontrollable muscle spasms and stiffness in the ankle during terminal stance (spasticity), as well as during transfers. In order to improve functional outcomes and further develop rehabilitation techniques, the underlying contributions of the corticospinal tract and spinal reflex circuit to ankle control needs to be better understood. Non-invasive tools that target the corticospinal and spinal reflex circuit are being used in clinical settings in order to improve functional outcomes in persons with spinal cord injury. Whole body vibration (WBV) is a non-invasive tool that has been shown to increase voluntary motor output and decrease spasticity in persons with spinal cord injury. These improvements in function may be due to changes in the corticospinal tract and spinal reflex circuits. In order to determine the relative contributions of the corticospinal tract and spinal reflex circuits to increased voluntary ankle control and decreased spasticity, we will measure changes in the corticospinal tract and spinal reflex excitability before and after a single session of vibration. We will then determine which change (corticospinal or spinal) contributes more to increased voluntary ankle control and decreased spasticity. This information will help guide future research to further improve walking ability in persons with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to consent and authorize use of Protected Health Information (PHI)
* Be between 18-85 years of age
* Be able to provide a letter of medical clearance for participation, if 70-85 years of age
* Have a SCI level of T12 of above, occurring more than 6 months ago
* Have a motor-incomplete severity classification (AIS C OR D)
* Have self-reported spasticity in at least one ankle
* Have a score of at least 2 indicating at least moderate spasticity on the Spinal Cord Assessment Tool for Spastic Reflexes (SCATS) clonus test in at least one ankle
* Have the ability to voluntarily move at least one ankle
* Must be able to stand and take at least 4 steps with or without assistive devices

Exclusion Criteria:

* Implanted metallic device in the head and/ or pacemaker
* Use of ankle-foot orthoses
* History of seizures
* History of frequent and/ or severe headaches
* Prior tendon or nerve transfer surgery
* Current pregnancy
* Inability or unwillingness to consent and Authorization for use of PHI
* Progressive or potentially progressive spinal lesions, including degenerative, or progressive vascular disorders of the spine and/or spinal cord
* Neurologic level below spinal level T12
* History of cardiovascular irregularities
* Problems with following instructions
* Orthopedic problems that would limit participation in the protocol (e.g. knee or hip flexion contractures of greater than 10 degrees).
* Active infection of any type, as infection may exacerbate spasticity resulting in inability to identify the influence of the treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Volitional Ankle Control-Tapping Task Performance | Through study completion at 2 weeks
  The participant will be seated with the foot positioned on a pressure sensitive switch embedded in a platform. Participants will be asked to voluntarily contract and relax the muscles that lift the front of the foot (while the heel stays in place on the platform) as quickly as possible for 10s for 4 trials with a 60s rest in between.
Ankle Spasticity-Ankle Clonus | Through study completion at 2 weeks
  This test measures the amount of spasticity in the ankle. Motion sensors to record the ankle joint angles will be used. For this test participants will sit upright. The leg will be raised and released allowing the front of the foot to land on the edge of a platform. The angle of the ankle and movement of the foot will be recorded as it drops and catches on the platform.

SECONDARY OUTCOMES:
Corticospinal tract excitability-Motor Evoked Potentials | Through study completion at 2 weeks
  This is a test to evaluate the connection between the brain and spinal cord. The skin over the muscles of the leg will be cleaned with an alcohol swab and a mildly abrasive paste (similar to the feel of toothpaste). Sensors that detect muscle activity will be placed over these sites. The location of these sensors will be marked on the skin at the beginning of each session using a non-toxic cosmetic pencil. Pulses of stimulation will be applied to the head using a type of non-invasive brain stimulation called transcranial magnetic stimulation (TMS). The strength of the stimulation will be increased until it causes the muscles of the leg to twitch, and the size of the muscle response will be recorded with the sensors placed over the muscles.
Low frequency depression | Through study completion at 2 weeks
  This test measures how the spinal cord responds to brief pulses of stimulation to the nerves of the legs. Recording electrodes will be taped to the muscles of the legs and brief pulses of stimulation will be applied to the legs.
Spinal Cord Assessment Tool for Spastic Reflexes | Through study completion at 2 weeks
  This test measures the amount of spasticity in the legs. A clinician will perform a series of 3 short tests commonly performed in the clinic to test the spasticity in the legs.
Ankle Isometric Strength Test | Through study completion at 2 weeks
  Test measures how strong the ankle muscles are. Participants will sit in a chair with foot pressed against a device that measures force. Participants will be asked to lift the front of the foot against the device as hard as possible.
Walking speed and walking pattern | Through study completion at 2 weeks
  This test measures how fast participants walk and the way the legs move during walking. Participants will wear sensors that track the position of the legs as they walk across the floor. They will be able to use whatever assistive devices they typically use (e.g., lower extremity orthotics, walker, forearm crutches).
Heart rate and %SpO2 | Through study completion at 2 weeks
  This test measures the heart rate of participants and the amount of oxygen in the blood. These 2 measures will be taken by placing a sensor on the finger, before and after each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Edelle Field-Fote, PT, PhD, Principal Investigator — Director of Spinal Cord Injury Research
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No